CLINICAL TRIAL: NCT05718609
Title: Efficacy of Quadruple Therapy Based on Fecal Molecular Antimicrobial Susceptibility Tests as First-line Treatment for Helicobacter Pylori Infection
Brief Title: Efficacy of Therapy Based on Fecal Molecular Antimicrobial Susceptibility Tests for Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1108
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-01

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Rabeprazole; Amoxicillin; Furazolidone; Clarithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Amoxicillin- and Clarithromycin-based BQT (Active Comparator): rabeprazole 10mg bid, amoxicillin 1g bid, clarithromycin 500mg bid, colloidal bismuth 200mg bid for 14 days
  Interventions: Drug: Rabeprazole; Drug: Colloidal Bismuth Pectin Granules; Drug: Amoxicillin; Drug: Clarithromycin
- Clarithromycin medication history-based BQT (Experimental): The clarithromycin medication history will be asked before the treatment and the therapy will be performed as follows: with clarithromycin medication history: rabeprazole 10mg bid, amoxicillin 1g bid, furazolidone 100mg bid, colloidal bismuth 200mg bid for 14 days; without clarithromycin medication history: rabeprazole 10mg bid, amoxicillin 1g bid, clarithromycin 500mg bid, colloidal bismuth 200mg bid for 14 days.
  Interventions: Drug: Rabeprazole; Drug: Colloidal Bismuth Pectin Granules; Drug: Amoxicillin; Drug: Furazolidone; Drug: Clarithromycin
- Antimicrobial susceptibility tests-based BQT (Experimental): Fecal molecular biology antimicrobial susceptibility tests will be performed before the treatment. The susceptibility of clarithromycin will be evaluated. The treatment regimen will be chosen according to the results of the antimicrobial susceptibility tests as follows: clarithromycin-sensitive: rabeprazole 10mg bid, amoxicillin 1g bid, clarithromycin 500mg bid, colloidal bismuth 200mg bid for 14 days; clarithromycin-resistant: rabeprazole 10mg bid, amoxicillin 1g bid, furazolidone 100mg bid, colloidal bismuth 200mg bid for 14 days.
  Interventions: Drug: Rabeprazole; Drug: Colloidal Bismuth Pectin Granules; Drug: Amoxicillin; Drug: Furazolidone; Drug: Clarithromycin

INTERVENTIONS:
Drug: Rabeprazole — proton-pump inhibitor (PPI)
Drug: Colloidal Bismuth Pectin Granules — Gastric mucosal protective drug with anti-H. pylori effect
Drug: Amoxicillin — Antibiotic for H. pylori eradication
Drug: Furazolidone — Antibiotic for H. pylori eradication
  Arms: Antimicrobial susceptibility tests-based BQT; Clarithromycin medication history-based BQT
Drug: Clarithromycin — Antibiotic for H. pylori eradication

SUMMARY:
This study aims to evaluate the efficacy and safety of 14-day quadruple therapy based on fecal molecular antimicrobial susceptibility tests for the first-line eradication of H. pylori infection, thus, providing more evidence to inform the value of fecal antimicrobial susceptibility tests in the first-line treatment of H. pylori infection.

DETAILED DESCRIPTION:
The eradication rate of H. pylori is decreasing year by year due to the occurrence of bacterial resistance, especially clarithromycin, one of the most widely-used antimicrobials against H. pylori. Understanding antibiotic resistance before treatment may be the main determinant of the successful eradication of H. pylori. Nevertheless, due to the invasive examination of sampling, the economy-benefit ratio, and the harsh cultivation conditions, traditional antimicrobial susceptibility test is rarely used before first-line eradication treatment in the real world. As an alternative, faster and simpler molecular methods applied to fecal samples obviate the need for endoscopy and provide the possibility to popularize the antimicrobial susceptibility tests catering to initial treatment. This study aims to explore the efficacy, safety, and economic benefits of the first-line therapy for H. pylori guided by fecal antimicrobial susceptibility tests.

ELIGIBILITY:
Inclusion Criteria:

Participants enrolled should meet the following criteria: (1) Participants aged 18-65 with no history of eradication treatment; (2) diagnosed as H. pylori infection by one or more of the following methodologies: gastric biopsy using histochemical staining, tissue culture, the 14C-urea breath test (UBT), the 13C-UBT, and/or fecal antigen; (3) were requested to undergo an endoscopy before the eradication treatment if they have alarm symptoms, a family history of gastric cancer or age over 40 years old without undergoing an endoscopy before; and (4) voluntarily participated in the clinical trial and have signed the informed consent.

Exclusion Criteria:

Potential participants will be screened on the following exclusion criteria: (1) Participants had a history of using antibiotics or bismuth within four weeks or acid inhibitor (including H2 receptor antagonist (H2RA), proton-pump inhibitor (PPI) or potassium-competitive acid blocker (P-CAB)) within two weeks before inclusion; (2) had an active peptic ulcer with complications such as hemorrhage, perforation, or obstruction; (3) had a history of esophagectomy or gastrectomy; (4) had an allergy to any study drug; (5) were pregnant or breastfeeding; (6) had a history of alcohol abuse or drug addiction; (7) existence of mental illness; or (8) without self-judgment ability.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori Eradication Rate | Six to eight weeks after completion of the medication
  Helicobacter pylori Eradication will be determined by 13C-urea breath test or 14C-urea breath test six to eight weeks after completion of the medication.

SECONDARY OUTCOMES:
Rate of Adverse Drug Reaction(ADR) | Within 7 days after completion of therapy
  Adverse drug reactions are classified into six types (with mnemonics): dose-related (Augmented), non-dose-related (Bizarre), dose-related and time-related (Chronic), time-related (Delayed), withdrawal (End of use), and failure of therapy (Failure).
Compliance Rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Du, Master, Study Chair — Second Affiliated Hospital of Zhejiang University, School of Medicine
Locations (1):
- Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
After the completion of this study, data are available upon reasonable request. Data are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD Sharing will be available from June 1st 2024.
Access Criteria: Data are available upon reasonable request. Data are available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Yu Z, Liu X, Qiao J, Shen W, Mao X, Lou G, Li Y, Xie Z, Ye J. Is Tailored Bismuth Quadruple Therapies (With Clarithromycin or Furazolidone) Based on Fecal Molecular Susceptibility Testing in First-Line Helicobacter pylori Eradication Treatment More Effective? A Three-Arm, Multicenter Randomized Clinical Trial. Helicobacter. 2025 Jan-Feb;30(1):e70018. doi: 10.1111/hel.70018. PMID 39924352
- [Derived] Wu Y, Wang Y, Liu X, Liao O, Lou G, Li Y, Wu H, Du Q, Ye J. Efficacy of quadruple therapy with clarithromycin based on faecal molecular antimicrobial susceptibility tests as first-line treatment for Helicobacter pylori infection: a protocol of a single-centre, single-blind, randomised clinical trial in China. BMJ Open. 2023 Jul 21;13(7):e072670. doi: 10.1136/bmjopen-2023-072670. PMID 37479526